CLINICAL TRIAL: NCT00935246
Title: Development of Escitalopram Genomic Device by Using Candidate Gene Approach and Genome-Wide Scanning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Principal Investigator, Doh Kwan Kim, M.D., Ph.D., Samsung Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008-12-042
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Depression; Continuous Antidepressant Abuse; Adverse Reaction to Drug
Keywords: Genomic devices; Prediction of Escitalopram Response; Depressed Patients
MeSH Terms: conditions — Depression; Drug-Related Side Effects and Adverse Reactions | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antidepressant treated group (Experimental): Antidepressant treated group: depressed patients treated with Escitalopram
  Interventions: Drug: Escitalopram
- other antidepressant treated group (No Intervention): other Antidepressant treated group: depressed patients treated with other antidepressant without escitalopram

INTERVENTIONS:
Drug: Escitalopram — Antidepressant administration of Escitalopram for 8 weeks under therapeutic dose
  Other Names: Escitalopram : Lexapro
  Arms: Antidepressant treated group

SUMMARY:
To reveal the genetic determinants of the treatment outcome of escitalopram in depressed patients (by using candidate gene approach and whole genome scanning).

DETAILED DESCRIPTION:
The purposes of this study are:

1. To reveal the genetic determinants of the treatment outcome of escitalopram in depressed patients (by using candidate gene approach and whole genome scanning)
2. To improve the success rate of escitalopram treatment response for depressed patients

ELIGIBILITY:
Inclusion Criteria:

1. Eligible patients were enrolled in the clinical trials program of hte Samsung Medical Center Geropsychiatry and Affective Disorder Clinics(Seoul, Korea). They received a semistructured diagnostic interview, the Samsung Psychiatric Evaluation Schedule. The affective disorder section of the Samsung Psychiatric Evaluation Schedule uses the Korean version of the structured clinical interview for the diagnostic and statistical manual of mental disorders, Fourth edition.
2. interview with one more patient's family member for objective diagnosis and final diagnosis decision by agreements of two more psychiatric physicians

Exclusion Criteria:

1. received psychotropic medication within 2 weeks of the study or fluoxetine within 4 weeks
2. potential study participants for pregnancy, significant medical conditions, abnormal laboratory baseline values, unstable psychiatric features(eg.suicidal), history of alcohol of drug dependence, seizures, head trauma with loss of consciousness, neurological illness, or concomitant Axis I psychiatric disorder.

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2008-12; Primary Completion 2011-10 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
antidepressant response at 2,4,6,8 weeks A/E monitoring at 1,2,4,6,8 weeks | 8 weeks

SECONDARY OUTCOMES:
biological value at 0 week and 8 weeks | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Doh Kwan Kim, PhD, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Kangnam, Seoul, South Korea